CLINICAL TRIAL: NCT04555174
Title: BIOTRONIK - SaFety and Performance Registry for an aLl-comers Subject Population With the Limus Eluting Orsiro Mission Stent System Within Daily Clinical Practice: BIOFLOW-VIII
Brief Title: BIOFLOW-VIII All-comers Orsiro Mission Safety and Performance Registry
Acronym: BIOFLOW-VIII
Status: Active, not recruiting | Type: Observational
Sponsor: Biotronik AG (Industry)
Collaborators: Biotronik France (Industry)
Responsible Party: Sponsor
Other Study IDs: C1902
Record Dates: First submitted 2020-09-02; First posted 2020-09-18 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia
Keywords: Observational registry; All-comers open-label registry; Percutaneous Coronary Intervention (PCI); Coronary revascularization; Orsiro Mission Drug Eluting Stent (DES); Stenting
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orsiro Mission DES: All subjects will be implanted with the Limus Eluting Orsiro Mission Stent System and followed up until 60 months.
  Interventions: Device: Orsiro Mission DES

INTERVENTIONS:
Device: Orsiro Mission DES — Percutaneous Coronary Intervention (PCI)

SUMMARY:
The BIOFLOW-VIII registry is a post-market clinical evaluation of the Orsiro Mission stent in subjects requiring coronary revascularization with Drug Eluting Stents (DES).

DETAILED DESCRIPTION:
BIOFLOW-VIII is a national, prospective, non-randomized, multi-center, open-label registry to confirm both, the acute performance as well as the mid- and long-term safety and clinical performance of the Orsiro Mission stent in an all-comers patient population within daily clinical practice.

A total of 868 subjects will be enrolled at approximately 50 study sites in France. Clinical follow-ups will take place at 6, 12, 36 and 60 months post index-procedure. Follow-ups can be conducted by telephone.

A subgroup analysis will evaluate the outcomes for patients treated ambulatory with same day discharge.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic coronary artery disease intended to be treated with an Orsiro Mission DES (silent ischemia is permitted)
* Subject has signed informed consent for data release
* Subject is geographically stable and willing to participate at all follow up assessments
* Subject is ≥ 18 years of age

Exclusion Criteria:

* Subject did not sign informed consent for data release
* Pregnancy
* Known allergy (which cannot be pre-treated) to all types of P2Y12 inhibitor (Clopidogrel, Ticagrelor, Prasugrel, Ticlopidine and Cangrelor; thus preventing the use of the appropriate P2Y12 inhibitor), aspirin, both heparin and bivalirudin, L-605 cobalt- chromium (Co-Cr) alloy or one of its major elements (cobalt, chromium, tungsten, nickel), silicon carbide, PLLA, mTOR inhibiting drugs such as sirolimus, or contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orsiro Mission is indicated for improving coronary luminal diameter in patients with symptomatic ischemic heart disease due to discrete de-novo stenotic lesions and in-stent restenotic lesions (length ≤ 40 mm) in the native coronary arteries with a reference vessel diameter of 2.25 mm to 4.0 mm.
Sampling Method: Non-Probability Sample
Enrollment: 872 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2027-02-19 (Estimated)

PRIMARY OUTCOMES:
Rate of Target Lesion Failure (TLF) at 12 months follow-up | 12 months
  TLF according to Academic Research Consortium-2 (ARC-2) definition: Composite of Cardiovascular Death, target-vessel Myocardial Infarction and clinically-driven Target Lesion Revascularization

SECONDARY OUTCOMES:
Rate of Target Lesion Failure (TLF) at 6, 36 and 60 months follow-up | 6, 36, and 60 months
Rate of Target Vessel Revascularization (TVR) at 6, 12, 36, and 60 months follow-up | 6, 12, 36, and 60 months
Rate of Target Lesion Revascularization (TLR) at 6, 12, 36, and 60 months follow-up | 6, 12, 36, and 60 months
Rate of Definite Stent Thrombosis at 6, 12, 36, and 60 months follow-up | 6, 12, 36, and 60 months
Percent of participants with Clinical Device Success defined as attainment of < 30% residual stenosis of the target lesion using Orsiro Mission only | Immediately after the intervention/procedure/surgery
Percent of participants with Clinical Procedural Success defined as attainment of < 30% residual stenosis of the target lesion using any percutaneous method without occurrence of in-hospital death, myocardial infarction or target lesion revascularization | From the intervention/procedure/surgery until hospital discharge, assessed up to 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul Barragan, MD, Principal Investigator — Polyclinique les Fleurs
Locations (41):
- France (41):
  - Clinique Esquirol Saint Hilaire, Agen
  - Clinique Axium, Aix-en-Provence
  - CH Antibes, Antibes
  - CH de Bastia, Bastia
  - GCS de cardiologie, Bayonne
  - Clinique Convert, Bourg-en-Bresse
  - Hôpital Privé Saint Martin, Caen
  - CHU de Cermont Ferrand, Clermont-Ferrand
  - CH Sud Francilien, Corbeil-Essonnes
  - CHU Henri Mondor, Créteil
  - Centre de cardiologie d'Evecquemont, Évecquemont
  - Clinique Mutualiste, Grenoble
  - CH d'Haguenau, Haguenau
  - Clinique Sainte Clotilde, La Réunion
  - Centre Hospitalier de La Rochelle, La Rochelle
  - Hôpital Louis Pasteur, Le Coudray
  - Hôpital Privé de l'Estuaire, Le Havre
  - Hôpital Marie Lannelongue, Le Plessis-Robinson
  - CH de Metz, Metz
  - Clinique Pont de Chaume, Montauban
  - Clinique du Millénaire, Montpellier
  - Clinique du Diaconat, Mulhouse
  - Hôpital Privé du Confluent, Nantes
  - Clinique Ambroise Paré, Neuilly-sur-Seine
  - Polyclinique Les Fleurs, Ollioules
  - Hôpital Lariboisière, Paris
  - Hôpital Saint Joseph, Paris
  - CH de Pau, Pau
  - Clinique La Croix du Sud, Quint-Fonsegrives
  - Polyclinique Saint Laurent, Rennes
  - Centre Cardiologique du Nord, Saint-Denis
  - Clinique Rhéna / GERC, Strasbourg
  - Nouvel Hopital Civil, Strasbourg
  - CH de Toulon, Toulon
  - CH de Tourcoing, Tourcoing
  - CHRU de Tours, Tours
  - Clinique Saint Joseph, Trélazé
  - CH de Valence, Valence
  - Polyclinique Vauban, Valenciennes
  - CH de Vannes, Vannes
  - Médpôle Lyon Villeurbanne, Villeurbanne

IPD SHARING:
Plan to Share IPD: No
The primary outcome data will be shared after publication of it.